CLINICAL TRIAL: NCT04248998
Title: Targeting Triple Negative BREAst Cancer Metabolism With a Combination of Chemotherapy and a Diet Mimicking FASTing Plus/Minus Metformin in the Preoperative Setting: the BREAKFAST Trial
Brief Title: Calorie Restriction With or Without Metformin in Triple Negative Breast Cancer
Acronym: BREAKFAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: IFOM ETS - The AIRC Institute of Molecular Oncology (Other); European Institute of Oncology (Other); University of Milan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 192/19; 2019-003093-13 (EudraCT Number)
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Triple-negative Breast Cancer
Keywords: Triple-negative breast cancer; Fasting-Mimicking Diet; Metformin; Tumor Metabolism; Cytotoxic Chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Metformin; AC protocol; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy plus Fasting-Mimicking Diet (FMD) (Experimental): Experimental Arm A will consist of 6 months of standard anthracycline-taxane preoperative chemotherapy in combination with triweekly cycles of 5-day FMD.
  Chemotherapy will consist of:
  * four triweekly cycles of doxorubicin 60 mg/mq plus cyclophosphamide 600 mg/mq, followed by
  * twelve consecutive cycles of weekly paclitaxel 80 mg/mq
  The FMD will consist of a triweekly 5-day regimen of a plant-based, calorie-restricted (600 KCal on day 1; 300 KCal on days 2-5), low-carbohydrate, low-protein diet. The FMD will be repeated up to a maximum of eight consecutive cycles.
  Interventions: Dietary Supplement: Fasting-mimicking diet; Drug: Preoperative chemotherapy
- Fasting-mimicking diet plus metformin plus chemotherapy (Experimental): Experimental Arm B will consist of 6 months of standard anthracycline-taxane preoperative chemotherapy in combination with triweekly cycles of 5-day FMD and daily metformin
  Chemotherapy will consist of:
  * four triweekly cycles of doxorubicin 60 mg/mq plus cyclophosphamide 600 mg/mq, followed by
  * twelve consecutive cycles of weekly paclitaxel 80 mg/mq
  The FMD will consist of a triweekly 5-day regimen of a plant-based, calorie-restricted (600 KCal on day 1; 300 KCal on days 2-5), low-carbohydrate, low-protein diet. The FMD will be repeated up to a maximum of eight consecutive cycles.
  Metformin will be administered at an initial dosage of 850 mg/dya, and then escalated to the maximum dosage of 1700/day (two 850 mg tablets) if well tolerated. Metformin will be interrupted 7 days before surgery.
  Interventions: Dietary Supplement: Fasting-mimicking diet; Drug: Metformin; Drug: Preoperative chemotherapy

INTERVENTIONS:
Dietary Supplement: Fasting-mimicking diet — Cyclic, 5-day, calorie-restricted (600 KCal on day 1; 300 KCal on days 2-5), low-carbohydrate, low protein diet every three weeks
Drug: Metformin — Metformin 850 mg twice a day
  Other Names: Metforal
  Arms: Fasting-mimicking diet plus metformin plus chemotherapy
Drug: Preoperative chemotherapy — Chemotherapy will consist of:
  * four triweekly cycles of doxorubicin 60 mg/mq plus cyclophosphamide 600 mg/mq, followed by
  * twelve consecutive cycles of weekly paclitaxel 80 mg/mq
  Other Names: doxorubicin+cyclophosphamide and paclitaxel

SUMMARY:
Glucose starvation and metformin have synergistic antitumor effects that are mediated through the concomitant inhibition of glycolysis and mitochondrial oxidative phosphorylation. The BREAKFAST trial will evaluate the antitumor activity of combining cyclic fasting-mimicking diet (FMD), which reproduces the in vitro effects of glucose starvation, plus/minus metformin with standard preperative anthracycline-taxane chemotherapy in patients with stage I-III TNBC

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is the most aggressive breast cancer subtype, and is associated with the lowest cure rates in the limited-stage disease setting, as well as with the lowest overall survival in the metastatic setting. Preclinical studies indicate that cycles of fasting or calorie-restricted, low-carbohydrate, low-protein diets, also known as fasting-mimicking diets (FMDs), have synergistic cytotoxic effects when combined with chemotherapy agents, such as doxorubicin or cisplatin, in several in vitro and in vivo tumor models, including murine TNBC models. More recently, intermittent fasting has demonstrated highly synergistic antitumor effects when combined with metformin; of note, these effects are mediated through the concomitant inhibition of glycolysis (via fasting-induced hypoglycemia) and metformin-induced inhibition of mitochondrial oxidative phosphorylation (OXPHOS). Finally, small reports published so far indicate that cyclic fasting and FMDs are well tolerated in cancer patients, and can be safety combined with standard antitumor treatments.

Based on these data, the BREAKFAST trial was designed to investigate the antitumor activity of cyclic FMD, alone or in combination with metformin, in patients with localized TNBC. In this study, 90 patients with stage I-III TNBC will be randomized in a 1:1 ratio to receive approximately 6 months of standard preoperative anthracycline plus taxane chemotherapy in combination with eight triweekly cycles of 5-day FMD (Arm A), or the same chemotherapy-FMD regimen plus daily metformin (Arm B). The primary objective of the study is to demonstrate that one or both experimental treatments increase the rate of pCR from 45% (historical data) to 65%

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study must meet all of the following criteria:

  1. Female sex
  2. Age ≥ 18 and ≤ 75 years.
  3. Evidence of a personally signed and dated informed consent document (ICD) indicating that the patient has been informed of all pertinent aspects of the study before enrollment
  4. Willingness and ability to comply with the prescribed FMD regimen, metformin intake, the scheduled visits, treatment plans, laboratory tests and other procedures.
  5. Histologically confirmed diagnosis of invasive TNBC candidate to neoadjuvant chemotherapy and subsequent curative surgery. On the basis of International Guidelines, TNBC is defined by absent or minimal (<1%) expression of oestrogen and progesterone receptors at IHC, and absence of HER2 over-expression or amplification, as defined as an IHC score of 0, 1+, or an IHC score of 2+ with in situ hybridization (ISH) analysis excluding HER2 gene amplification.
  6. Patients with localized disease (clinical stage I-III according to TNM). Patients with Stage I TNBC will be included only if the primary tumor is at least 10 mm in greatest dimension (clinical T1c as determined through baseline MRI assessment).
  7. Presence of an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
  8. Presence of adequate bone marrow and organ function as defined by the following laboratory values:

     1. ANC ≥ 1.5 x 103/l
     2. platelets ≥ 100 x 103/l
     3. hemoglobin ≥ 9.0 g/dl
     4. calcium (corrected for serum albumin) within normal limits or ≤ grade 1 according to NCI-CTCAE version 5.0 if not clinically significant
     5. potassium within the normal limits, or corrected with supplements
     6. creatinine < 1.5 ULN
     7. blood uric acid < 10 mg/dl
     8. ALT and AST ≤ 2 x ULN
     9. total bilirubin < 1.5 ULN except for patients with Gilbert syndrome who may only be included if the total bilirubin is < 3.0 x ULN or direct bilirubin < 1.5 x ULN
     10. Fasting glucose ≤ 250 mg/dl.
  9. Female patients of childbearing potential must agree to sexual abstinence or to use two highly effective methods of contraception throughout the study and for at least six months after the end of the FMD. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide. A patient is of childbearing potential if, in the opinion of the Investigator, she is biologically capable of having children and is sexually active.
  10. Female patients are not of childbearing potential if they meet at least one of the following criteria:

      1. Have undergone a documented hysterectomy and/or bilateral oophorectomy
      2. Have medically confirmed ovarian failure
      3. Achieved post-menopausal status, defined as: ≥ 12 months of non-therapy-induced amenorrhea or surgically sterile (absence of ovaries) and have a serum FSH level within the laboratory's reference range for postmenopausal females.

Exclusion Criteria:

* Patients eligible for this study must not meet any of the following criteria:

  1. Prior systemic treatment for breast cancer or other malignancies within 5 years of treatment enrollment.
  2. Prior treatment with anthracyclines
  3. Diagnosis of other malignancies in advanced stages (unresectable, locally advanced or metastatic), or that required systemic (neo)adjuvant chemotherapy in the previous 5 years. Other malignancies diagnosed more than 5 years before the diagnosis of breast cancer must have been radically treated without evidence of relapse at the moment of patient enrollment in the trial.
  4. Body mass index (BMI) < 20 kg/m2.
  5. History of alcohol abuse.
  6. Non-intentional weight loss ≥ 5% in the previous 3 months, unless the patient has a BMI > 22 kg/m2 and weight loss has been lower than 10% at the time of enrollment in the study; or non-intentional weight loss of ≥ 10% in the previous 3 months, unless the patients has a BMI > 25 kg/m2 and weight loss has been lower than 15% at the time of the enrollment in the study. In both cases, weight must have been stable for at least one month before study enrollment.
  7. Active pregnancy or breast feeding.
  8. Known active B or C hepatitis or human immunodeficiency virus (HIV) infection, or occasional finding of active hepatitis B/C infection during screening tests before chemotherapy initiation, as defined as positive polymerase chain reaction (PCR) testing for HBV-DNA and HCV-RNA and qualitative PCR for HIV-RNA, or requiring active treatment at study enrollment.
  9. Serious infections in the previous 4 weeks before the FMD initiation, including, but not limited to, potential hospitalizations for complications of infections, bacteriemia or serious pneumonitis.
  10. Active autoimmune diseases requiring systemic treatments (e.g. systemic steroids or immune suppressants).
  11. Active chronic therapy with systemic steroids at a dose ≥ 10 mg per day of prednisone or equivalent at study enrollment.
  12. Known recent diagnosis of hypothyroidism requiring systemic replacement hormonal therapy and without stabilization of hormonal profile (fT3, fT4 and TSH within the normal range).
  13. Diagnosis of type 1 or 2 diabetes mellitus requiring pharmacologic therapy (including, but not limited to, insulin, secretagogues and metformin). A diagnosis of type 2 diabetes mellitus not requiring pharmacological treatments based on the judgment of a diabetologist, is compatible with patient enrollment in the trial.
  14. Active gastric or intestinal ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small intestine resection.
  15. Anamnesis of clinically significant heart disease including:

      1. angina pectoris, coronary bypass, symptomatic pericarditis, myocardial infarction in the previous 12 months from the beginning of experimental therapy;
      2. congestive heart failure (NYHA III-IV).
  16. Anamnesis of clinically meaningful cardiac arrhythmias, such as ventricular tachycardia, chronic atrial fibrillation, complete bundle branch block, high grade atrio-ventricular block like bi-fascicular block, type II Mobitz and third grade atrio-ventricular block, nodal arrhythmias, supra-ventricular arrhythmia.
  17. Left ventricular ejection fraction lower than 50% at the cardiac scan with radionuclides or at echocardiography.
  18. Previous episodes of symptomatic hypotension leading to loss of consciousness.
  19. Baseline plasma fasting glucose ≤ 60 mg/dL.
  20. Medical or psychiatric comorbidities rendering the patient not candidate to the clinical trial, according to the investigator's judgement.
  21. Other cardiac, liver, lung or renal comorbidities, not specified in the previous inclusion or exclusion criteria, but potentially exposing the patient to a high risk of lactic acidosis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 36 months
  Rate of pathologic complete responses (pCRs)

SECONDARY OUTCOMES:
Severe adverse events | 36 months
  Incidence of severe (grade 3 or 4) adverse events according to CTCAE v 5.0
Safety of the experimental treatments | 36 months
  Incidence of treatment-related adverse events (AEs)
Compliance with the experimental treatment | 36 months
  Patients' ability to adhere to the prescribed FMD regimen and pharmacological treatment according to the analysis of daily food diaries and diaries related to metformin intake
RFS | 60 months
  Relapse-free survival
DMFS | 60 months
  Distant metastasis-free survival
OS | 60 months
  Overall Survival
Short-term modifications of plasma glycemia (mg/dl) | 30 months
  Short-term modifications of plasma glucose levels, as defined as changes in peripheral blood venous plasma glucose concentration before and after each FMD cycle
Long-term modifications of plasma glycemia (mg/dl) | 30 months
  Long-term modifications of plasma glucose concentration, as defined as changes in peripheral blood venous plasma glucose concentration measured before consecutive FMD cycles
Short-term modifications of serum insulin concentration (µU/ml) | 30 months
  Short-term modifications of serum insulin concentration, as defined as changes in peripheral blood venous serum insulin concentration before and after each FMD cycle
Long-term modifications of serum insulin concentration (µU/ml) | 30 months
  Long-term modifications of serum insulin concentration, as defined as changes in peripheral blood venous serum insulin concentration measured before consecutive FMD cycles
Short-term modifications of serum IGF-1 concentration (ng/ml) | 30 months
  Short-term modifications of serum IGF-1 concentration, as defined as changes in peripheral blood venous serum IGF-1 concentration before and after each FMD cycle
Long-term modifications ofserum IGF-1 concentration (ng/ml) | 30 months
  Long-term modifications of blood IGF-1 concentration, as defined as changes in serum IGF-1 concentration measured before consecutive FMD cycles
Short-term modifications of blood lipid profile by UPLC-MS and HPLC-ELDS | 30 months
  Short-term modifications of blood lipid profile, as defined as changes in plasma lipids before and after individual FMD cycles
Long-term modifications of blood lipid profile by UPLC-MS and HPLC-ELDS | 30 months
  Long-term modifications of blood lipid profile, as defined as changes in plasma lipids assessed before consecutive FMD cycles
Clinical tumor response | 30 months
  To estimate clinical tumor responses, as assessed through Magnetic Resonance Imaging (MRI) evaluations according to RECIST 1.1 criteria before surgery
Gene expression profiles | 36 months
  To correlate baseline metabolic gene expression, as assessed through RNA-seq analysis, with patient probability to achieve a pCR. In particular, the expression of genes encoding for catalytic, regulatory and scaffolding subunits of PP2A will be evaluated.
Mutational analyses | 36 months
  To correlate mutational tumor profiles, as assessed through whole-genome sequencing analysis, with patient probability to achieve a pCR. In particular, the expression of genes encoding for catalytic, regulatory and scaffolding subunits of PP2A will be evaluated.
Short-term modifications of plasma amino acid profile by UPLC-QDa Mass detector system (Waters) | 30 months
  Short-term modifications of plasma amino acid profile, as defined as changes in plasma amino acids before and after individual FMD cycles
Long-term modifications of plasma amino acid profile by UPLC-QDa Mass detector system (Waters) | 30 months
  Long-term modifications of plasma amino acid profile, as defined as changes in plasma amino acids assessed before consecutive FMD cycles

CONTACTS AND LOCATIONS:
Overall Officials: Filippo de Braud, Professor, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Claudio Vernieri, M.D. PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Ferlay J, Colombet M, Soerjomataram I, Dyba T, Randi G, Bettio M, Gavin A, Visser O, Bray F. Cancer incidence and mortality patterns in Europe: Estimates for 40 countries and 25 major cancers in 2018. Eur J Cancer. 2018 Nov;103:356-387. doi: 10.1016/j.ejca.2018.07.005. Epub 2018 Aug 9. PMID 30100160
- [Result] Iqbal J, Ginsburg O, Rochon PA, Sun P, Narod SA. Differences in breast cancer stage at diagnosis and cancer-specific survival by race and ethnicity in the United States. JAMA. 2015 Jan 13;313(2):165-73. doi: 10.1001/jama.2014.17322. PMID 25585328
- [Result] Kassam F, Enright K, Dent R, Dranitsaris G, Myers J, Flynn C, Fralick M, Kumar R, Clemons M. Survival outcomes for patients with metastatic triple-negative breast cancer: implications for clinical practice and trial design. Clin Breast Cancer. 2009 Feb;9(1):29-33. doi: 10.3816/CBC.2009.n.005. PMID 19299237
- [Result] Gobbini E, Ezzalfani M, Dieras V, Bachelot T, Brain E, Debled M, Jacot W, Mouret-Reynier MA, Goncalves A, Dalenc F, Patsouris A, Ferrero JM, Levy C, Lorgis V, Vanlemmens L, Lefeuvre-Plesse C, Mathoulin-Pelissier S, Petit T, Uwer L, Jouannaud C, Leheurteur M, Lacroix-Triki M, Cleaud AL, Robain M, Courtinard C, Cailliot C, Perol D, Delaloge S. Time trends of overall survival among metastatic breast cancer patients in the real-life ESME cohort. Eur J Cancer. 2018 Jun;96:17-24. doi: 10.1016/j.ejca.2018.03.015. Epub 2018 Apr 13. PMID 29660596
- [Result] Park S, Koo JS, Kim MS, Park HS, Lee JS, Lee JS, Kim SI, Park BW. Characteristics and outcomes according to molecular subtypes of breast cancer as classified by a panel of four biomarkers using immunohistochemistry. Breast. 2012 Feb;21(1):50-7. doi: 10.1016/j.breast.2011.07.008. Epub 2011 Aug 23. PMID 21865043
- [Result] Lehmann BD, Bauer JA, Chen X, Sanders ME, Chakravarthy AB, Shyr Y, Pietenpol JA. Identification of human triple-negative breast cancer subtypes and preclinical models for selection of targeted therapies. J Clin Invest. 2011 Jul;121(7):2750-67. doi: 10.1172/JCI45014. PMID 21633166
- [Result] Schmid P, Adams S, Rugo HS, Schneeweiss A, Barrios CH, Iwata H, Dieras V, Hegg R, Im SA, Shaw Wright G, Henschel V, Molinero L, Chui SY, Funke R, Husain A, Winer EP, Loi S, Emens LA; IMpassion130 Trial Investigators. Atezolizumab and Nab-Paclitaxel in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2018 Nov 29;379(22):2108-2121. doi: 10.1056/NEJMoa1809615. Epub 2018 Oct 20. PMID 30345906
- [Result] Sharma P, Lopez-Tarruella S, Garcia-Saenz JA, Khan QJ, Gomez HL, Prat A, Moreno F, Jerez-Gilarranz Y, Barnadas A, Picornell AC, Monte-Millan MD, Gonzalez-Rivera M, Massarrah T, Pelaez-Lorenzo B, Palomero MI, Gonzalez Del Val R, Cortes J, Fuentes-Rivera H, Morales DB, Marquez-Rodas I, Perou CM, Lehn C, Wang YY, Klemp JR, Mammen JV, Wagner JL, Amin AL, O'Dea AP, Heldstab J, Jensen RA, Kimler BF, Godwin AK, Martin M. Pathological Response and Survival in Triple-Negative Breast Cancer Following Neoadjuvant Carboplatin plus Docetaxel. Clin Cancer Res. 2018 Dec 1;24(23):5820-5829. doi: 10.1158/1078-0432.CCR-18-0585. Epub 2018 Jul 30. PMID 30061361
- [Result] Tutt A, Tovey H, Cheang MCU, Kernaghan S, Kilburn L, Gazinska P, Owen J, Abraham J, Barrett S, Barrett-Lee P, Brown R, Chan S, Dowsett M, Flanagan JM, Fox L, Grigoriadis A, Gutin A, Harper-Wynne C, Hatton MQ, Hoadley KA, Parikh J, Parker P, Perou CM, Roylance R, Shah V, Shaw A, Smith IE, Timms KM, Wardley AM, Wilson G, Gillett C, Lanchbury JS, Ashworth A, Rahman N, Harries M, Ellis P, Pinder SE, Bliss JM. Carboplatin in BRCA1/2-mutated and triple-negative breast cancer BRCAness subgroups: the TNT Trial. Nat Med. 2018 May;24(5):628-637. doi: 10.1038/s41591-018-0009-7. Epub 2018 Apr 30. PMID 29713086
- [Result] O'Shaughnessy J, Schwartzberg L, Danso MA, Miller KD, Rugo HS, Neubauer M, Robert N, Hellerstedt B, Saleh M, Richards P, Specht JM, Yardley DA, Carlson RW, Finn RS, Charpentier E, Garcia-Ribas I, Winer EP. Phase III study of iniparib plus gemcitabine and carboplatin versus gemcitabine and carboplatin in patients with metastatic triple-negative breast cancer. J Clin Oncol. 2014 Dec 1;32(34):3840-7. doi: 10.1200/JCO.2014.55.2984. Epub 2014 Oct 27. PMID 25349301
- [Result] Rugo HS, Barry WT, Moreno-Aspitia A, Lyss AP, Cirrincione C, Leung E, Mayer EL, Naughton M, Toppmeyer D, Carey LA, Perez EA, Hudis C, Winer EP. Randomized Phase III Trial of Paclitaxel Once Per Week Compared With Nanoparticle Albumin-Bound Nab-Paclitaxel Once Per Week or Ixabepilone With Bevacizumab As First-Line Chemotherapy for Locally Recurrent or Metastatic Breast Cancer: CALGB 40502/NCCTG N063H (Alliance). J Clin Oncol. 2015 Jul 20;33(21):2361-9. doi: 10.1200/JCO.2014.59.5298. Epub 2015 Jun 8. PMID 26056183
- [Result] Yardley DA, Coleman R, Conte P, Cortes J, Brufsky A, Shtivelband M, Young R, Bengala C, Ali H, Eakel J, Schneeweiss A, de la Cruz-Merino L, Wilks S, O'Shaughnessy J, Gluck S, Li H, Miller J, Barton D, Harbeck N; tnAcity investigators. nab-Paclitaxel plus carboplatin or gemcitabine versus gemcitabine plus carboplatin as first-line treatment of patients with triple-negative metastatic breast cancer: results from the tnAcity trial. Ann Oncol. 2018 Aug 1;29(8):1763-1770. doi: 10.1093/annonc/mdy201. PMID 29878040
- [Result] Carey LA, Dees EC, Sawyer L, Gatti L, Moore DT, Collichio F, Ollila DW, Sartor CI, Graham ML, Perou CM. The triple negative paradox: primary tumor chemosensitivity of breast cancer subtypes. Clin Cancer Res. 2007 Apr 15;13(8):2329-34. doi: 10.1158/1078-0432.CCR-06-1109. PMID 17438091
- [Result] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986
- [Result] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Result] Poggio F, Bruzzone M, Ceppi M, Ponde NF, La Valle G, Del Mastro L, de Azambuja E, Lambertini M. Platinum-based neoadjuvant chemotherapy in triple-negative breast cancer: a systematic review and meta-analysis. Ann Oncol. 2018 Jul 1;29(7):1497-1508. doi: 10.1093/annonc/mdy127. PMID 29873695
- [Result] Loibl S, O'Shaughnessy J, Untch M, Sikov WM, Rugo HS, McKee MD, Huober J, Golshan M, von Minckwitz G, Maag D, Sullivan D, Wolmark N, McIntyre K, Ponce Lorenzo JJ, Metzger Filho O, Rastogi P, Symmans WF, Liu X, Geyer CE Jr. Addition of the PARP inhibitor veliparib plus carboplatin or carboplatin alone to standard neoadjuvant chemotherapy in triple-negative breast cancer (BrighTNess): a randomised, phase 3 trial. Lancet Oncol. 2018 Apr;19(4):497-509. doi: 10.1016/S1470-2045(18)30111-6. Epub 2018 Feb 28. PMID 29501363
- [Result] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Result] McAndrew N, DeMichele A. Neoadjuvant Chemotherapy Considerations in Triple-Negative Breast Cancer. J Target Ther Cancer. 2018 Feb;7(1):52-69. Epub 2018 Feb 14. PMID 29577076
- [Result] Houvenaeghel G, Goncalves A, Classe JM, Garbay JR, Giard S, Charytensky H, Cohen M, Belichard C, Faure C, Uzan S, Hudry D, Azuar P, Villet R, Gimbergues P, Tunon de Lara C, Martino M, Lambaudie E, Coutant C, Dravet F, Chauvet MP, Chereau Ewald E, Penault-Llorca F, Esterni B. Characteristics and clinical outcome of T1 breast cancer: a multicenter retrospective cohort study. Ann Oncol. 2014 Mar;25(3):623-628. doi: 10.1093/annonc/mdt532. Epub 2014 Jan 7. PMID 24399079
- [Result] Vernieri C, Casola S, Foiani M, Pietrantonio F, de Braud F, Longo V. Targeting Cancer Metabolism: Dietary and Pharmacologic Interventions. Cancer Discov. 2016 Dec;6(12):1315-1333. doi: 10.1158/2159-8290.CD-16-0615. Epub 2016 Nov 21. PMID 27872127
- [Result] Lee C, Raffaghello L, Brandhorst S, Safdie FM, Bianchi G, Martin-Montalvo A, Pistoia V, Wei M, Hwang S, Merlino A, Emionite L, de Cabo R, Longo VD. Fasting cycles retard growth of tumors and sensitize a range of cancer cell types to chemotherapy. Sci Transl Med. 2012 Mar 7;4(124):124ra27. doi: 10.1126/scitranslmed.3003293. Epub 2012 Feb 8. PMID 22323820
- [Result] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Result] de Groot S, Vreeswijk MP, Welters MJ, Gravesteijn G, Boei JJ, Jochems A, Houtsma D, Putter H, van der Hoeven JJ, Nortier JW, Pijl H, Kroep JR. The effects of short-term fasting on tolerance to (neo) adjuvant chemotherapy in HER2-negative breast cancer patients: a randomized pilot study. BMC Cancer. 2015 Oct 5;15:652. doi: 10.1186/s12885-015-1663-5. PMID 26438237
- [Result] Dorff TB, Groshen S, Garcia A, Shah M, Tsao-Wei D, Pham H, Cheng CW, Brandhorst S, Cohen P, Wei M, Longo V, Quinn DI. Safety and feasibility of fasting in combination with platinum-based chemotherapy. BMC Cancer. 2016 Jun 10;16:360. doi: 10.1186/s12885-016-2370-6. PMID 27282289
- [Result] Braghiroli MI, de Celis Ferrari AC, Pfiffer TE, Alex AK, Nebuloni D, Carneiro AS, Caparelli F, Senna L, Lobo J, Hoff PM, Riechelmann RP. Phase II trial of metformin and paclitaxel for patients with gemcitabine-refractory advanced adenocarcinoma of the pancreas. Ecancermedicalscience. 2015 Aug 11;9:563. doi: 10.3332/ecancer.2015.563. eCollection 2015. PMID 26316884
- [Result] Martin-Castillo B, Pernas S, Dorca J, Alvarez I, Martinez S, Perez-Garcia JM, Batista-Lopez N, Rodriguez-Sanchez CA, Amillano K, Dominguez S, Luque M, Stradella A, Morilla I, Vinas G, Cortes J, Cuyas E, Verdura S, Fernandez-Ochoa A, Fernandez-Arroyo S, Segura-Carretero A, Joven J, Perez E, Bosch N, Garcia M, Lopez-Bonet E, Saidani S, Buxo M, Menendez JA. A phase 2 trial of neoadjuvant metformin in combination with trastuzumab and chemotherapy in women with early HER2-positive breast cancer: the METTEN study. Oncotarget. 2018 Nov 2;9(86):35687-35704. doi: 10.18632/oncotarget.26286. eCollection 2018 Nov 2. PMID 30479698
- [Result] Tsakiridis T, Hu C, Skinner HD, et al. Initial reporting of NRG-LU001 (NCT02186847), randomized phase II trial of concurrent chemoradiotherapy (CRT) +/- metformin in locally advanced Non-Small Cell Lung Cancer (NSCLC). Journal of Clinical Oncology. 2019;37(15_suppl):8502-8502.
- [Result] Jiralerspong S, Palla SL, Giordano SH, Meric-Bernstam F, Liedtke C, Barnett CM, Hsu L, Hung MC, Hortobagyi GN, Gonzalez-Angulo AM. Metformin and pathologic complete responses to neoadjuvant chemotherapy in diabetic patients with breast cancer. J Clin Oncol. 2009 Jul 10;27(20):3297-302. doi: 10.1200/JCO.2009.19.6410. Epub 2009 Jun 1. PMID 19487376
- [Result] Masuda N, Lee SJ, Ohtani S, Im YH, Lee ES, Yokota I, Kuroi K, Im SA, Park BW, Kim SB, Yanagita Y, Ohno S, Takao S, Aogi K, Iwata H, Jeong J, Kim A, Park KH, Sasano H, Ohashi Y, Toi M. Adjuvant Capecitabine for Breast Cancer after Preoperative Chemotherapy. N Engl J Med. 2017 Jun 1;376(22):2147-2159. doi: 10.1056/NEJMoa1612645. PMID 28564564
- [Result] Hammond ME, Hayes DF, Dowsett M, Allred DC, Hagerty KL, Badve S, Fitzgibbons PL, Francis G, Goldstein NS, Hayes M, Hicks DG, Lester S, Love R, Mangu PB, McShane L, Miller K, Osborne CK, Paik S, Perlmutter J, Rhodes A, Sasano H, Schwartz JN, Sweep FC, Taube S, Torlakovic EE, Valenstein P, Viale G, Visscher D, Wheeler T, Williams RB, Wittliff JL, Wolff AC; American Society of Clinical Oncology; College of American Pathologists. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer (unabridged version). Arch Pathol Lab Med. 2010 Jul;134(7):e48-72. doi: 10.5858/134.7.e48. PMID 20586616
- [Result] Wolff AC, Hammond MEH, Allison KH, Harvey BE, Mangu PB, Bartlett JMS, Bilous M, Ellis IO, Fitzgibbons P, Hanna W, Jenkins RB, Press MF, Spears PA, Vance GH, Viale G, McShane LM, Dowsett M. Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer: American Society of Clinical Oncology/College of American Pathologists Clinical Practice Guideline Focused Update. Arch Pathol Lab Med. 2018 Nov;142(11):1364-1382. doi: 10.5858/arpa.2018-0902-SA. Epub 2018 May 30. PMID 29846104
- [Result] Sardanelli F, Boetes C, Borisch B, Decker T, Federico M, Gilbert FJ, Helbich T, Heywang-Kobrunner SH, Kaiser WA, Kerin MJ, Mansel RE, Marotti L, Martincich L, Mauriac L, Meijers-Heijboer H, Orecchia R, Panizza P, Ponti A, Purushotham AD, Regitnig P, Del Turco MR, Thibault F, Wilson R. Magnetic resonance imaging of the breast: recommendations from the EUSOMA working group. Eur J Cancer. 2010 May;46(8):1296-316. doi: 10.1016/j.ejca.2010.02.015. Epub 2010 Mar 19. PMID 20304629
- [Result] Kuhl C. The current status of breast MR imaging. Part I. Choice of technique, image interpretation, diagnostic accuracy, and transfer to clinical practice. Radiology. 2007 Aug;244(2):356-78. doi: 10.1148/radiol.2442051620. PMID 17641361
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Oktay K, Harvey BE, Partridge AH, Quinn GP, Reinecke J, Taylor HS, Wallace WH, Wang ET, Loren AW. Fertility Preservation in Patients With Cancer: ASCO Clinical Practice Guideline Update. J Clin Oncol. 2018 Jul 1;36(19):1994-2001. doi: 10.1200/JCO.2018.78.1914. Epub 2018 Apr 5. PMID 29620997
- [Result] Hammond ME, Hayes DF, Dowsett M, Allred DC, Hagerty KL, Badve S, Fitzgibbons PL, Francis G, Goldstein NS, Hayes M, Hicks DG, Lester S, Love R, Mangu PB, McShane L, Miller K, Osborne CK, Paik S, Perlmutter J, Rhodes A, Sasano H, Schwartz JN, Sweep FC, Taube S, Torlakovic EE, Valenstein P, Viale G, Visscher D, Wheeler T, Williams RB, Wittliff JL, Wolff AC. American Society of Clinical Oncology/College Of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer. J Clin Oncol. 2010 Jun 1;28(16):2784-95. doi: 10.1200/JCO.2009.25.6529. Epub 2010 Apr 19. PMID 20404251
- [Result] Wolff AC, Hammond MEH, Allison KH, Harvey BE, Mangu PB, Bartlett JMS, Bilous M, Ellis IO, Fitzgibbons P, Hanna W, Jenkins RB, Press MF, Spears PA, Vance GH, Viale G, McShane LM, Dowsett M. Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer: American Society of Clinical Oncology/College of American Pathologists Clinical Practice Guideline Focused Update. J Clin Oncol. 2018 Jul 10;36(20):2105-2122. doi: 10.1200/JCO.2018.77.8738. Epub 2018 May 30. PMID 29846122
- [Result] Carey LA, Metzger R, Dees EC, Collichio F, Sartor CI, Ollila DW, Klauber-DeMore N, Halle J, Sawyer L, Moore DT, Graham ML. American Joint Committee on Cancer tumor-node-metastasis stage after neoadjuvant chemotherapy and breast cancer outcome. J Natl Cancer Inst. 2005 Aug 3;97(15):1137-42. doi: 10.1093/jnci/dji206. PMID 16077072
- [Result] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Derived] Ligorio F, Vingiani A, Torelli T, Sposetti C, Drufuca L, Iannelli F, Zanenga L, Depretto C, Folli S, Scaperrotta G, Capri G, Bianchi GV, Ferraris C, Martelli G, Maugeri I, Provenzano L, Nichetti F, Agnelli L, Lobefaro R, Fuca G, Fotia G, Mariani L, Morelli D, Ladisa V, De Santis MC, Lozza L, Trecate G, Belfiore A, Brich S, Bertolotti A, Lorenzini D, Ficchi A, Martinetti A, Sottotetti E, Arata A, Corsetto P, Sorrentino L, Rediti M, Salvadori G, Minucci S, Foiani M, Apolone G, Pagani M, Pruneri G, de Braud F, Vernieri C. Early downmodulation of tumor glycolysis predicts response to fasting-mimicking diet in triple-negative breast cancer patients. Cell Metab. 2025 Feb 4;37(2):330-344.e7. doi: 10.1016/j.cmet.2024.11.004. Epub 2024 Dec 17. PMID 39694040